CLINICAL TRIAL: NCT05995678
Title: A Mixed Methods Pilot Trial of the STEP Home Workshop to Improve Reintegration and Reduce Suicide Risk for Recently Transitioned Veterans
Acronym: SH-SP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D4535-R
Record Dates: First submitted 2023-06-20; First posted 2023-08-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: TBI; Suicide Prevention; Veterans; PTSD; Transdiagnostic; Anger
Keywords: Veterans; TBI; Transdiagnostic; Intervention; Suicide Prevention; PTSD; Reintegration
MeSH Terms: conditions — Suicide Prevention; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Following T1 baseline assessment, participants will be randomized to STEP-Home-SP + Usual Care or Usual Care (UC) using randomly permuted block sizes stratified by presence or absence of SI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEP-Home-SP + Usual Care (Experimental): The core skills of emotional regulation and problem solving are introduced and integrated throughout all Veteran-specific reintegration content modules for practice and repetition for 12 weeks. Attention training augments emotional regulation and problem solving core skills and is interspersed throughout group and individual sessions. Additional 30-minute individual skill building and goal setting sessions occur ~4-6 times based on individual Veteran needs
  Interventions: Behavioral: STEP-Home-SP; Behavioral: Transition Assistance Program; Behavioral: VA Solid Start
- Usual Care (Active Comparator): UC will include the Transition Assistance Program (TAP) as scheduled by DOD prior to military separation, VA Solid Start post-separation, and educational augmentation post-separation.
  Interventions: Behavioral: Transition Assistance Program; Behavioral: VA Solid Start

INTERVENTIONS:
Behavioral: STEP-Home-SP — This group will meet for ~1.5 hours/week for 12 weeks. The core skills of Emotional Regulation (ER) and Problem Solving (PS) are introduced and then integrated throughout all Veteran-specific content modules for practice and repetition for 12 weeks. Attention training augments ER and PS skills and is interspersed throughout the group and individual sessions. Additional 30-minute individual skills building and goal setting sessions occur up to 6 times based on individual Veteran needs. STEP-Home staff will work in pairs to run workshops per established protocols. Workshops will be conducted via VA approved video telehealth.
  Arms: STEP-Home-SP + Usual Care
Behavioral: Transition Assistance Program — Provides training, skills, and information to help transitioning service members and their families prepare for the military to civilian transition. Each service member works with a TAP counselor to identify needs and post transition goals to build an Individual Transition Plan, in addition to TAP core curriculum courses.
  Other Names: TAP
Behavioral: VA Solid Start — VA Solid Start includes a series of outreach calls and emails to all Veterans at 90-, 180-, and 365-days post service separation. Callers follow a standard script to describe services available through VA and provide contact information for desired services.

SUMMARY:
Risk of Veteran suicide is elevated during the first year of transition from military service to civilian life. Most Veteran suicides occur among Veterans who are not connected to VA healthcare. Suicide prevention and connection to care are therefore critical for recently transitioning Veterans. Transitioning Veterans require services to provide them with suicide prevention education, skills to manage their transition effectively, and support in their access to VA healthcare. Convenient, accessible, palatable, patient-centered care options that are cost-effective, easy to implement nationwide, and target domains known to mitigate suicide risk are needed during this critical transition period. This proposal would bridge this important healthcare gap using STEP-Home-SP, a transdiagnostic, non-stigmatizing, skills-based workshop. STEP-Home-SP will provide Veterans with suicide prevention education, skills to improve transition, support to access VA care, and a platform to decrease social isolation early in their military to civilian transition, thereby reducing suicide risk downstream.

DETAILED DESCRIPTION:
Veterans face a "deadly gap" during their first year of transition from military to civilian life with limited available psychiatric services and increased suicide risk factors. During this critical transition period, Veteran suicide rate is double that of active service members and the general Veteran population. An average of 20 Veterans die from suicide each day, but only 6 of the 20 use VA services. VA care engagement has been shown to mitigate suicide risk; therefore, promoting engagement during the "deadly gap" could be essential to suicide prevention. Transitioning Veterans require outreach and services to provide them with support in their access to VA healthcare, suicide prevention education, and skills to manage their transition effectively. This proposal would bridge this important healthcare gap using STEP-Home. STEP-Home is an evidence-based, transdiagnostic, video telehealth rehabilitation workshop to improve reintegration, social support, and functioning among Veterans with high clinical comorbidity. STEP-Home is non-clinical, cost-effective, and skills-focused to maximally engage Veterans not participating in treatment who may be resistant to traditional "mental health" diagnostically focused approaches. To date, STEP-Home has not been adapted for the unique needs of recently transitioning Veterans or augmented for suicide prevention. This proposal will adapt and refine STEP-Home specifically for recently transitioning Veterans and add suicide prevention content and skills to create STEP-Home-SP. The proposed pilot study is designed to support STEP-Home and suicide prevention content experts in their refinement and evaluation of STEP-Home-SP. The investigators will utilize the VA/Department of Defense Identity Repository (VADIR) to recruit recently transitioned Veterans nationwide. In Aim 1, the investigators will develop STEP-Home-SP by adapting the STEP-Home telehealth intervention to specifically target recently transitioned Veterans and augment the workshop to include suicide prevention. In Aim 2, the investigators will conduct a two-arm proof-of-concept acceptability and feasibility randomized controlled trial (RCT) of STEP-Home-SP versus Enhanced Usual Care (EUC=current standard of care + educational packet on suicide risk and connection to VA care) in recently transitioned Veterans. Lastly, the investigators will explore reintegration status, VA care initiation, and candidate outcomes for STEP-Home-SP relative to EUC to inform a future full-scale RCT. If successful, fostering social, vocational, and community connection; building emotion regulation and impulse control skills; facilitating safety planning; and providing education and access to VA care upstream should result in decreased suicide risk during this critical transition and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Recently transitioned Veterans within one year of separation from military service
* Self-reported functional impairment or reintegration difficulties as measured by the Military-to-Civilian Questionnaire (any item score > 1 indicating "some difficulty"; M2CQ; [71])
* Sufficient English fluency
* Agree to participate (informed consent/HIPAA)

Exclusion Criteria:

* Active psychosis
* Imminent or acute high suicide risk requiring immediate crisis intervention (low-moderate non-imminent risk for suicide is allowed)
* Current moderate or severe substance use disorder
* Neurological diagnosis excluding TBI

  * Participants with mild substance use disorder will be allowed
  * Substance use is a common behavior that may contribute to reintegration difficulties and suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility- recruitment interest | Through study completion, an average of one year.
  ratio interested of those approached for the workshop
Feasibility- enrollment | Through study completion, an average of one year.
  Ratio enrolled (consented) of those approached, greater than 20% of those interested enroll in the proposed time frame
Feasibility- qualitative via Narrative Evaluation of Intervention Interview | Through study completion, an average of 3 months.
  Identification of challenges and facilitators during the recruitment process as assessed by study staff as well as feedback from focus group participants generated using the Narrative Evaluation of Intervention Interview (NEII). This is an interview composed of 16 open ended questions that allows participants to evaluate the process and outcomes of the intervention. Reviewers will generate a list of themes based on the responses to this interview.
Feasibility- Treatment Fidelity/adherence | Through study completion, an average of 1 week.
  Supervisor and therapist Likert rating of adherence to content for core skills and treatment modules, less than 20% deviations on a treatment fidelity scale. Lower scores indicate stronger treatment fidelity, with each question being answered on a scale from 1 (Strongly Agree) to 5 (Strongly Disagree).
Acceptability- Veteran adherence | Through study completion, an average of one year.
  Attendance rate for the 12-session workshop
Acceptability- Quantitative satisfaction via Client satisfaction questionnaire Change | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Client satisfaction questionnaire (CSQ-8), total scores range from 8 to 32 with higher scores indicating higher satisfaction. A priori criteria is that greater than 80% of participants will score greater that a 24 on the CSQ-8.
Reintegration status- Military to Civilian Questionnaire (M2CQ) Change | Assessed at screening, baseline (0 weeks), T4 (after 12 weeks) and T5 (after 24 weeks)
  16 questions are answered on a scale from 0 (no difficulty) to 4 (extreme difficulty), with lower scores indicating more successful reintegration.

SECONDARY OUTCOMES:
Engagement in VA Care | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Electronic medical record data (if available) showing occurrence of one or more healthcare appointments

OTHER OUTCOMES:
Difficulties in Emotional Regulation Scale (DERS) | Assessed at baseline (0 weeks), T2 (after 4 weeks), T3 (after 8 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  36 statements are each ranked on the following scale by participants: 1 almost never (0-10%), 2 sometimes (11-35%), 3 about half the time (36-55%), 4 most of the time (66-90%), or 5 almost always (91-100%). This produces scores for 6 subscales: nonacceptance of emotional responses; difficulty engaging in goal-directed behavior; impulse control difficulties; lack of emotional awareness; limited access to emotion regulation strategies; lack of emotional clarity.
Problem Solving Inventory (PSI) | Assessed at baseline (0 weeks), T2 (after 4 weeks), T3 (after 8 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants rank 35 statements on a Likert scale from 1 (strongly agree) to 6 (strongly disagree). This generates a total score and 3 subscale scores for the following categories: Approach Avoidance, Personal Control, and Problem Solving Confidence.
Attention-Related Cognitive Errors Scale (ARCES) | Assessed at baseline (0 weeks), T2 (after 4 weeks), T3 (after 8 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  12 questions are ranked on a Likert Scale from 1 (never) to 5 (very often) with higher scores indicating more frequent attention related cognitive errors.
Suicidal Ideation- The Columbia-Suicide Severity Rating Scale (C-SSRS) | Assessed at screening, baseline (0 weeks), T2 (after 4 weeks), T3 (after 8 weeks), T4 (after 12 weeks), and T5 (after 24 weeks). Will also be administered as needed following workshop sessions.
  Participants are asked 5 questions designed to assess severity of suicide risk. Questions are answered yes or no, with endorsement of active suicidal ideation with intent being considered high risk and suicidal ideation without intent considered moderate risk.
Post-deployment Readjustment Inventory (PDRI) | Assessed at screening, baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  36 statements are ranked by participants on a scale from 1 (not at all) to 5 (extremely). Total score is calculated by the sum of each of the subscales: Career, Health, Intimate relationships, social readjustment, concerns about deployment, and PTSD symptoms. Higher scores indicate less successful post-deployment readjustment.
State-Trait Anger Expression Inventory (STAXI-2) | Assessed at screening, baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Measures the experience, expression, and control of anger. Participants rank each of the statements on a scale of 1 (not at all) to 4 (very much so) for section 1 and 1 (almost never) to 4 (almost always) for sections 2 and 3. Higher scores indicate high experience/expression and low control of anger.
Functional status measured using the WHO Disability Assessment Schedule 2.0 12-item (WHODAS-2.0) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants indicate how much difficulty they have had in the last 30 days for each of the statements on the assessment on a scale from 0 (none) to 4 (Extreme/cannot do). Higher scores indicate greater levels of disability.
Stigma- Perceived Barriers to Care Survey | Assessed at baseline (0 weeks), T2 (after 4 weeks), T3 (after 8 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants rank each of the survey items on the scale from 1 (strongly agree) to 5 (strongly disagree) with lower scores indicating that the item is a greater barrier to care.
Quality of Life Scale (QOLS) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants answer each question on a 7 point scale. It is scored by adding up the score on each item to get a minimum potential score of 16 and a maximum total score of 112. Higher scores indicate a higher quality of life.
Psychosocial Functioning- The Brief Inventory of Psychosocial Functioning (IPF-Brief) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants rank each of the 7 statements based on their overall experience over the past month on a scale from 0 (not at all) to 6 (very much). 7 is marked if the statement is not applicable. Higher scores indicate more impaired psychosocial functioning.
Social support subscale of the Deployment Risk and Resilience Inventory (DRRI-2) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants rank each of the ten questions from this subscale on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree) and total subscale score is calculated by adding up the responses from each of the questions. Lower scores indicate lower levels of social support.
Interpersonal Needs Questionnaire (INQ) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Each of the 15 questions are answered on a scale from 1 (Not at all true for me) to 7 (very true for me). 6 out of the 15 questions are reverse coded. Higher scores indicate that more interpersonal needs are not met.
Depression- Patient Health Questionnaire (PHQ-9) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants rank 9 questions on a scale from 0 (not at all) to 3 (Nearly every day) based on how often in the last 2 weeks they have been bothered by the problems listed. Then they rate the severity of the difficulty any problems they have experienced are causing on a scale from "not difficult at all" to "extremely difficult." Higher scores indicate higher depression severity.
Hopelessness- Beck Hopelessness Scale | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants answer 20 true or false questions that are scored based on an answer key. Answers that indicate hopelessness are added up, with higher scores indicating higher levels of hopelessness/pessimism.
Self-injurious thoughts and behaviors interview (SITBI) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  This interview asks a wide variety of questions related to suicidal ideations, plans, gestures, attempts, and non-suicidal self injurious behaviors. There are 72 possible questions, but some are only asked if a specific behavior is endorsed. Higher scores indicate higher levels of thoughts and feelings related to suicide and self-injurious behaviors.
Suicide Coping/Safety Behaviors- Suicide Related Coping Scale (SRCS) | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Participants answer 17 questions on a 5 point Likert scale from 0-4 (Strongly Disagree to Strongly Agree). Total score is determined by reverse scoring negatively worded items and then summing the items. Higher scores indicate better coping skills.
Gateway to vocational and community activities- Treatment & Activities Survey | Assessed at baseline (0 weeks), T4 (after 12 weeks), and T5 (after 24 weeks)
  Treatment & Activities Survey developed by STEP-Home staff asks participants to list the types of treatment (psychotherapy, medication, group therapy) that they have participated in within the last month, what they receive the treatment for, and whether it is administered by the VA or outside of the VA. Participants also answer if they have participated in other activities in the last month (school, work, community, etc.) and whether those activities are at or outside of the VA.
Kessler-6 brief mental health screen | Baseline (0 weeks)
  The Kessler Psychological Distress Scale (K6) is a 6 item measure of participants' emotional state. Questions are scored from 0 (none of the time) to 4 (all of the time) with a minimum score of 0 and a maximum score of 24. Higher scores indicate higher levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B Fortier, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No additional IPD will be shared besides the deidentified/anonymized data set and data dictionary will be shared.